CLINICAL TRIAL: NCT01465542
Title: Treatment of Acetaminophen Toxicity With Intravenous vs. Oral N-acetylcysteine: A Retrospective Review
Brief Title: Treatment of APAP Toxicity With IV and Oral NAC 2008-2011
Status: Completed | Type: Observational
Sponsor: Akron Children's Hospital (Other)
Responsible Party: Principal Investigator, Martha Blackford, PharmD, PharmD, Akron Children's Hospital
Other Study IDs: APAP & NAC 2008-2011
Record Dates: First submitted 2011-10-31; First posted 2011-11-04 (Estimated); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Acetaminophen Toxicity
Keywords: Acetaminophen Toxicity; Acetaminophen Overdose; N-acetylcysteine; Liver Toxicity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Oral NAC: Patients receiving oral NAC treatment after an acute acetaminophen ingestion.
- IV NAC: Patients receiving IV NAC after an acute Acetaminophen ingestion.

SUMMARY:
Retrospective chart review of patients who receive N-acetylcysteine for Acetaminophen(APAP) toxicity to assess length of oral vs. IV treatment and the effect of a Clinical Pharmacology and Toxicology division in the management of APAP ingestions.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to CHMCA between June 1, 2008 to June 30, 2011
* Qualifying ICD-9 diagnosis code for the following APAP overdose situations: poisoning, accidental, suicide attempt, therapeutic use, assault, and undetermined (965.4, E850.4, E950.0, E935.4, E962.0, E980.0)
* Serum APAP concentration above the possible hepatotoxic line on the Rumack-Matthew's nomogram if obtained > 4 hours post ingestion
* Between ages 0-21 years on date of admission
* Acute APAP ingestion

Exclusion Criteria:

* Serum APAP concentrations not actually documented
* Did not receive the oral or IV NAC treatment
* Preexisting liver disease such as cirrhosis or hepatitis C
* Patient > 21 years of age on the date of admission
* Chronic APAP ingestion

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric and adolescent patients with acetaminophen toxicity.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2011-06; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Length of NAC treatment in hours | Retrospective data collection for patient's hospital admission, max estimated 5days
  Length of NAC treatment (in hours) for both IV and PO formulations used in patients with APAP toxicity

SECONDARY OUTCOMES:
Pharmacology & Toxicology consults | Retrospective data collection for length of patient's hospital admission, max estimated 5 days
  Documenting whether or not a pharmacology & toxicology consult was obtained during the patient's hospital admission for APAP toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Martha Blackford, PharmD, Principal Investigator — CHMCA
Locations (1):
- Children's Hospital Medical Center of Akron, Akron, Ohio, United States

REFERENCES:
- [Background] Dart RC, Erdman AR, Olson KR, Christianson G, Manoguerra AS, Chyka PA, Caravati EM, Wax PM, Keyes DC, Woolf AD, Scharman EJ, Booze LL, Troutman WG; American Association of Poison Control Centers. Acetaminophen poisoning: an evidence-based consensus guideline for out-of-hospital management. Clin Toxicol (Phila). 2006;44(1):1-18. doi: 10.1080/15563650500394571. PMID 16496488
- [Background] Kanter MZ. Comparison of oral and i.v. acetylcysteine in the treatment of acetaminophen poisoning. Am J Health Syst Pharm. 2006 Oct 1;63(19):1821-7. doi: 10.2146/ajhp060050. PMID 16990628
- [Background] Whyte IM, Francis B, Dawson AH. Safety and efficacy of intravenous N-acetylcysteine for acetaminophen overdose: analysis of the Hunter Area Toxicology Service (HATS) database. Curr Med Res Opin. 2007 Oct;23(10):2359-68. doi: 10.1185/030079907X219715. PMID 17705945
- [Background] Yarema MC, Johnson DW, Berlin RJ, Sivilotti ML, Nettel-Aguirre A, Brant RF, Spyker DA, Bailey B, Chalut D, Lee JS, Plint AC, Purssell RA, Rutledge T, Seviour CA, Stiell IG, Thompson M, Tyberg J, Dart RC, Rumack BH. Comparison of the 20-hour intravenous and 72-hour oral acetylcysteine protocols for the treatment of acute acetaminophen poisoning. Ann Emerg Med. 2009 Oct;54(4):606-14. doi: 10.1016/j.annemergmed.2009.05.010. Epub 2009 Jun 25. PMID 19556028